CLINICAL TRIAL: NCT03368066
Title: Is Adrenal Insufficiency Under-diagnosed in Hospitalized Cirrhosis Patients?
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Zachary Henry, MD, Principal Investigator, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20212
Record Dates: First submitted 2017-11-20; First posted 2017-12-11 (Actual); Results first posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Adrenal Insufficiency; Cirrhosis; Spur Cell Anemia; Lecithin Acyltransferase Deficiency
MeSH Terms: conditions — Adrenal Insufficiency; Fibrosis; Abetalipoproteinemia; Lecithin Cholesterol Acyltransferase Deficiency | interventions — Cosyntropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Hospitalized cirrhosis patients (Experimental): Administration of cortisol stimulation test to assess for presence or absence of adrenal insufficiency
  Interventions: Drug: Cosyntropin

INTERVENTIONS:
Drug: Cosyntropin — Administer 250mcg cosyntropin to hospitalized cirrhosis patients to assess for the presence of adrenal insufficiency

SUMMARY:
The hepatoadrenal syndrome has been well described in the literature and is known to be associated with poorer outcomes in both stable and critically ill cirrhotic patients. In chronic liver disease, adrenal (and more specifically cortisol) insufficiency is thought to be a byproduct of altered lipid metabolism that results in decreased HDL production and thus decreased delivery of cholesterol to the adrenal for subsequent corticosteroid production. Studies to date have implicated lecithin-cholesterol acetyltransferase (LCAT) as the key enzyme which is deficient in some cirrhotic patients, leading to an impaired ability to esterify cholesterol and thus a loss of normal cellular functioning and membrane stability. The investigators seek to quantify this LCAT deficiency in a cohort of cirrhotic patients and demonstrate its association with various abnormal physiologies associated with chronic liver disease, including spur cell anemia, low HDL levels, and adrenal insufficiency.

Hospitalized cirrhotic patients at UVA that meet study eligibility criteria will be approached by a member of the study team to obtain consent for participation. If a patient agrees to become a study subject, they will have an approximate total of 35ml of blood drawn the following morning. Lab tests to be performed include: peripheral blood smear, lipid panel, free cortisol, cortisol binding globulin, serum cholesterol esters (surrogate for LCAT enzyme activity), and a standard-dose cortisol stimulation test. The latter involves blood drawn with the initial collection, administration of an intravenous 250mcg dose of synthetic ACTH, and then repeat small-volume blood draws at 30 minutes and 60 minutes later.

Subjects will be classified as adrenally sufficient or insufficient on the basis of as standard-dose cortisol stimulation test. Variables of interest for comparison between the groups include MELD score, Child-Turcotte-Pugh (CTP) classification, high-density lipoprotein (HDL) levels, presence of spur cell anemia, serum cholesterol ester percentage (surrogate for LCAT enzymatic activity), cortisol binding globulin levels, and free cortisol levels. Student's t-test and Chi Square tests will be utilized to determine significance; a p <0.05 value will be used as our threshold for significance. If multiple factors are found to be significantly different in a univariate fashion between classification groups, a multivariate logistic regression analysis will be performed for adjusted analysis. The investigators will also seek to define any correlations between variables. Furthermore, the investigators will assess correlation between MELD score and serum cholesterol ester percentage, spur cell anemia, HDL levels, cortisol binding globulin levels, and free cortisol levels; similar correlate analysis will be done using CTP classification instead of MELD score.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years
* Diagnosis of cirrhosis
* Admission to hospital

Exclusion Criteria:

* Age < 18 years
* Prior enrollment in study (i.e. readmission)
* Prisoner
* Pregnancy
* Prednisone or Hydrocortisone use in last 24 hours

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2019-03-12 (Actual); Study Completion 2019-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Henry, MD, Principal Investigator — University of Virginia School of Medicine, Department of Medicine, Division of Gastroenterology & Hepatology
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fede G, Spadaro L, Tomaselli T, Privitera G, Germani G, Tsochatzis E, Thomas M, Bouloux PM, Burroughs AK, Purrello F. Adrenocortical dysfunction in liver disease: a systematic review. Hepatology. 2012 Apr;55(4):1282-91. doi: 10.1002/hep.25573. PMID 22234976
- [Background] O'Beirne J, Holmes M, Agarwal B, Bouloux P, Shaw S, Patch D, Burroughs A. Adrenal insufficiency in liver disease - what is the evidence? J Hepatol. 2007 Sep;47(3):418-23. doi: 10.1016/j.jhep.2007.06.008. Epub 2007 Jun 28. PMID 17629587
- [Background] Triantos CK, Marzigie M, Fede G, Michalaki M, Giannakopoulou D, Thomopoulos K, Garcovich M, Kalafateli M, Chronis A, Kyriazopoulou V, Jelastopoulou E, Nikolopoulou V, O'Beirne J, Burroughs AK. Critical illness-related corticosteroid insufficiency in patients with cirrhosis and variceal bleeding. Clin Gastroenterol Hepatol. 2011 Jul;9(7):595-601. doi: 10.1016/j.cgh.2011.03.033. Epub 2011 Apr 8. PMID 21545846
- [Background] Fede G, Spadaro L, Tomaselli T, Privitera G, Piro S, Rabuazzo AM, Sigalas A, Xirouchakis E, O'Beirne J, Garcovich M, Tsochatzis E, Purrello F, Burroughs AK. Assessment of adrenocortical reserve in stable patients with cirrhosis. J Hepatol. 2011 Feb;54(2):243-50. doi: 10.1016/j.jhep.2010.06.034. Epub 2010 Sep 15. PMID 21056503
- [Background] Fede G, Spadaro L, Tomaselli T, Privitera G, Scicali R, Vasianopoulou P, Thalassinos E, Martin N, Thomas M, Purrello F, Burroughs AK. Comparison of total cortisol, free cortisol, and surrogate markers of free cortisol in diagnosis of adrenal insufficiency in patients with stable cirrhosis. Clin Gastroenterol Hepatol. 2014 Mar;12(3):504-12.e8; quiz e23-4. doi: 10.1016/j.cgh.2013.08.028. Epub 2013 Aug 24. PMID 23978347
- [Background] Tan T, Chang L, Woodward A, McWhinney B, Galligan J, Macdonald GA, Cohen J, Venkatesh B. Characterising adrenal function using directly measured plasma free cortisol in stable severe liver disease. J Hepatol. 2010 Nov;53(5):841-8. doi: 10.1016/j.jhep.2010.05.020. Epub 2010 Jul 17. PMID 20739086
- [Background] Jang JY, Kim TY, Sohn JH, Lee TH, Jeong SW, Park EJ, Lee SH, Kim SG, Kim YS, Kim HS, Kim BS. Relative adrenal insufficiency in chronic liver disease: its prevalence and effects on long-term mortality. Aliment Pharmacol Ther. 2014 Oct;40(7):819-26. doi: 10.1111/apt.12891. Epub 2014 Jul 30. PMID 25078874
- [Background] Tamer S, Cefle K, Palanduz S, Vatansever S. Rheological properties of blood in patients with chronic liver disease. Clin Hemorheol Microcirc. 2002;26(1):9-14. PMID 11904466
- [Background] Tamer S, Cefle K, Gokkusu C, Ademoglu E, Ozturk S, Vatansever S, Palanduz S, Guler K. Comparison of rheological parameters in patients with post hepatitic and alcoholic cirrhosis. Clin Hemorheol Microcirc. 2007;36(3):247-52. PMID 17361026
- [Background] Kakimoto H, Imai Y, Kawata S, Inada M, Ito T, Matsuzawa Y. Altered lipid composition and differential changes in activities of membrane-bound enzymes of erythrocytes in hepatic cirrhosis. Metabolism. 1995 Jul;44(7):825-32. doi: 10.1016/0026-0495(95)90233-3. PMID 7616839
- [Background] Alexopoulou A, Vasilieva L, Kanellopoulou T, Pouriki S, Soultati A, Dourakis SP. Presence of spur cells as a highly predictive factor of mortality in patients with cirrhosis. J Gastroenterol Hepatol. 2014 Apr;29(4):830-4. doi: 10.1111/jgh.12473. PMID 24325340
- [Background] Cooper RA, Diloy Puray M, Lando P, Greenverg MS. An analysis of lipoproteins, bile acids, and red cell membranes associated with target cells and spur cells in patients with liver disease. J Clin Invest. 1972 Dec;51(12):3182-92. doi: 10.1172/JCI107145. PMID 4640953
- [Background] Miller JP. Dyslipoproteinaemia of liver disease. Baillieres Clin Endocrinol Metab. 1990 Dec;4(4):807-32. doi: 10.1016/s0950-351x(05)80080-1. PMID 2082907
- [Background] Kaiser T, Kinny-Koster B, Bartels M, Berg T, Scholz M, Engelmann C, Seehofer D, Becker S, Ceglarek U, Thiery J. Cholesterol esterification in plasma as a biomarker for liver function and prediction of mortality. BMC Gastroenterol. 2017 Apr 20;17(1):57. doi: 10.1186/s12876-017-0614-9. PMID 28427335

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 patients were excluded - 1 patient did not undergo cortisol stimulation testing due to administrative error and 4 patients had compensated cirrhosis (Child Pugh A).
Groups:
- Normal Adrenal Response: Delta cortisol response to 250mcg Cosyntropin > 9 micrograms/dL
- Relative Adrenal Insufficiency: Delta cortisol response to 250mcg Cosyntropin < 9 micrograms/dL
Period: Overall Study
Arm/Group | Normal Adrenal Response | Relative Adrenal Insufficiency
Started | 58 | 37
Completed | 58 | 37
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Hospitalized Cirrhosis Patients
Number analyzed (Participants) | 95
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [52 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 56
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 95
Etiology of Cirrhosis [Count of Participants; unit: Participants] — If a patient had more than one etiology of cirrhosis (i.e. Alcohol and Hepatitis C) or an etiology of cirrhosis not otherwise categorized separately (i.e. autoimmune hepatitis, hemochromatosis, etc.), they were captured in the "other" category.
  Participants
    Alcohol | 33
    Non-alcoholic steatohepatitis | 22
    Hepatitis C | 9
    Cryptogenic | 14
    Other | 17
Decompensation [Count of Participants; unit: Participants]
  Ascites | 88
  Hepatic Encephalopathy | 55
  Esophageal Varices | 68
Hepatocellular Carcinoma [Count of Participants; unit: Participants] | 11
Aldosterone Antagonist Use [Count of Participants; unit: Participants] | 55
Beta Blocker Use [Count of Participants; unit: Participants] | 38
Midodrine Use [Count of Participants; unit: Participants] | 6
Infection During Hospitalization [Count of Participants; unit: Participants] | 24
Intensive Care Unit Stay During Hospitalization [Count of Participants; unit: Participants] | 8
Acute Kidney Injury (AKI) [Count of Participants; unit: Participants] — Acute kidney injury (AKI) was defined by the Kidney Disease Improving Global Outcomes (KDIGO) criteria:
  Stage 1: increase in creatinine 1.5-1.9 times baseline within 7 days or increase in creatinine >= 0.3 mg/dL within 48 hours or urine volume <0.5ml/kg/h for 6-12 hours.
  Stage 2: increase in creatinine 2-2.9 times baseline within 7 days or urine volume <0.5ml/kg/h for >= 12 hours.
  Stage 3: increase in creatinine >= 3.0 times baseline within 7 days or creatinine >= 4.0 or initiation of renal replacement therapy or urine volume <0.3ml/kg/h for >= 24 hours or anuria >= 12 hours.
  Participants
    Stage 1 | 24
    Stage 2 | 2
    Stage 3 | 4
Mean Arterial Pressure [Median (Inter-Quartile Range); unit: mmHg] | 78 [72 to 85]
Sodium [Median (Inter-Quartile Range); unit: mEq/L] | 136 [132 to 138]
Potassium [Median (Inter-Quartile Range); unit: mEq/L] | 3.9 [3.6 to 4.5]
Model for End-Stage Liver Disease (MELD) score [Median (Inter-Quartile Range); unit: units on a scale] — The MELD Score ranges from 6 to 40, with a score of 6 reflecting none to minimal loss of liver + renal function and 40 reflecting severe liver and/or renal impairment.
  units on a scale | 17 [13 to 21]
Child Pugh classification [Count of Participants; unit: Participants] — The Child-Pugh classification is a well-known classification system that characterizes severity of liver disease and is associated with increasing mortality as the classification increases. 5 variables are used in classifying a patient - degree of ascites, degree of hepatic encephalopathy, bilirubin level, albumin level, and the prothrombin time (or internationalized normal ratio). Class A is mild/compensated disease, Class B is decompensated disease, and Class C is severely decompensated disease.
  Participants
    B | 51
    C | 44
Albumin [Median (Inter-Quartile Range); unit: g/dL] | 2.8 [2.4 to 3.0]
HDL [Median (Inter-Quartile Range); unit: mg/dL] | 23 [12 to 34]
Baseline Cortisol [Median (Inter-Quartile Range); unit: micrograms/dL] | 7.9 [5.0 to 11.0]
Delta Cortisol [Median (Inter-Quartile Range); unit: micrograms/dL] | 10.0 [7.6 to 12.7]
Free Cortisol [Median (Inter-Quartile Range); unit: micrograms/dL] | 0.6 [0.3 to 1.0]
Cortisol Binding Globulin [Median (Inter-Quartile Range); unit: mg/dL] | 1.7 [1.4 to 2.2]
Cholesterol Esters [Median (Inter-Quartile Range); unit: percentage of esterified cholesterol] | 66 [60 to 69]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Cholesterol Esterification Deficiency
Description: A percent quantification of serum cholesterol esterification will be measured via blood draw. Low values represent deficiency in esterification, which is a surrogate measure of lecthicin-cholesterol acetyltransferase (LCAT) enzymatic deficiency.
Time Frame: 24 hours
Population: 2 patients in normal adrenal response group and 3 patients in RAI group were missing cholesterol ester percentage measurements
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Adrenal Response | Relative Adrenal Insufficiency
Number analyzed (Participants) | 56 | 34
Participants | 10 | 11

2. Primary Outcome: Number of Participants With Spur Cell Anemia
Description: A peripheral blood smear will be obtained and assessed for presence of acanthocytes (spur cells). Spur cell anemia is defined as a serum hemoglobin < 10g/dL and the presence of >= 5% spur cells on blood smear.
Time Frame: 24 hours
Population: 2 patients with RAI were missing peripheral smears to assess for the presence of spur cells
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Adrenal Response | Relative Adrenal Insufficiency
Number analyzed (Participants) | 58 | 35
Participants | 6 | 8

3. Primary Outcome: Participant Transplant-Free Survival
Description: Transplant and Death are considered equivalent outcomes
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Adrenal Response | Relative Adrenal Insufficiency
Number analyzed (Participants) | 58 | 37
Participants | 41 | 16

4. Secondary Outcome: Number of Participants With Relative Adrenal Insufficiency (RAI)
Description: A baseline total cortisol level will be obtained and then patients will receive a standard-dose synthetic ACTH (250mcg of Cosyntropin) stimulation test to assess for the presence of adrenal insufficiency. RAI is defined as a change in the total cortisol level in response to the stimulation test of <9mcg/dL when measured 60 minutes after the Cosyntropin is administered.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Hospitalized Cirrhosis Patients
Number analyzed (Participants) | 95
Participants | 37

5. Secondary Outcome: Number of Participants With Low Free Cortisol
Description: Patients will have their free cortisol levels measured to assess for deficiency.
Time Frame: 24 hours
Population: 1 patient from normal adrenal response group was missing free cortisol data
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Adrenal Response | Relative Adrenal Insufficiency
Number analyzed (Participants) | 57 | 37
Participants | 6 | 1

6. Secondary Outcome: Number of Participants Who Received Liver Transplantation at 90 Days
Description: Patients who received a liver transplant within 90 days of enrollment
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Adrenal Response | Relative Adrenal Insufficiency
Number analyzed (Participants) | 58 | 37
Participants | 6 | 5

7. Secondary Outcome: Number of Participants Who Received Liver Transplantation at 6 Months
Description: Patients who received a liver transplant within 6 months of enrollment
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Adrenal Response | Relative Adrenal Insufficiency
Number analyzed (Participants) | 58 | 37
Participants | 8 | 6

8. Secondary Outcome: Number of Participants Who Died Within Index Hospitalization
Description: Patients who died within the same hospitalization as enrollment
Time Frame: Within Hospitalization
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Adrenal Response | Relative Adrenal Insufficiency
Number analyzed (Participants) | 58 | 37
Participants | 1 | 1

9. Secondary Outcome: Number of Participants Who Died at 30 Days
Description: Patients who died within 30 days of enrollment
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Adrenal Response | Relative Adrenal Insufficiency
Number analyzed (Participants) | 58 | 37
Participants | 4 | 4

10. Secondary Outcome: Number of Participants Who Died at 90 Days
Description: Patients who died within 90 days of enrollment
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Adrenal Response | Relative Adrenal Insufficiency
Number analyzed (Participants) | 58 | 37
Participants | 5 | 12

11. Secondary Outcome: Number of Participants Who Died at 6 Months
Description: Patients who died within 6 months of enrollment
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Adrenal Response | Relative Adrenal Insufficiency
Number analyzed (Participants) | 58 | 37
Participants | 9 | 15

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Hospitalized Cirrhosis Patients
All-Cause Mortality (participants affected / at risk) | 25/100
Serious Adverse Events (participants affected / at risk) | 25/100
Other Adverse Events (participants affected / at risk) | 1/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hospitalized Cirrhosis Patients (N=100)
Liver-related death (Hepatobiliary disorders) | 24 (24) — Death partially or completely attributed to patient's liver disease
Non-liver-related death (General disorders) | 1 (1) — Death not related to underlying liver disease
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hospitalized Cirrhosis Patients (N=100)
Nausea (Gastrointestinal disorders) | 1 (1) — Patient who experienced nausea after Cosyntropin administration, resolved with IV anti-emetic therapy

LIMITATIONS AND CAVEATS:
Excluded patients with Child Pugh A (compensated cirrhosis) given low number (4).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT03368066/Prot_SAP_000.pdf